CLINICAL TRIAL: NCT06162780
Title: The Efficacy and Safety of TEER for Severe DMR Patients of Low to Intermediate Surgery Risk (TESLA-R)--a Multi-center, Prospective Cohort Study
Brief Title: TEER for Severe DMR of Low to Intermediate Surgery Risk
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Peking University Shenzhen Hospital (Other); Dongguan People's Hospital (Other Government); First People's Hospital of Foshan (Other); The Second People's Hospital of Foshan (Other); The First Affiliate Hospital of Guangxi Medical College (Unknown); Affiliated Hospital of Guangdong Medical University (Other); Huizhou Third People's Hospital (Unknown); Jiangmen Central Hospital (Other); Guangzhou Panyu Center Hospital (Unknown); Meizhou People's Hospital (Other); Suzhou Municipal Hospital (Other); The General Hospital of Southern Theater Command (Other); People's Hospital of Nanhai District, Foshan (Unknown); Nanfang Hosptial, China (Unknown); Southern Medical University, China (Other); First Affiliated Hospital of Shantou University Medical College (Other); Shantou Central Hospital (Other); Sichuan Provincial People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Yueyang Central Hospital (Other); ZhuZhou Central Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Central South University Xiangya Hospital (Unknown); Zhongshan People's Hospital, Guangdong, China (Other); Foshan Fosun Chancheng Hospital (Unknown)
Responsible Party: Principal Investigator, Yangxin Chen, Chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2023-1019-03
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Mitral Regurgitation
Keywords: degenerative mitral regurgitation; transcatheter mitral valve edge-to-edge repair; surgery risk
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TEER group: Severe DMR patients of low to intermediate surgery risk who underwent TEER.
  Interventions: Diagnostic Test: ultrasonic cardiography (UCG); Procedure: TEER

INTERVENTIONS:
Diagnostic Test: ultrasonic cardiography (UCG) — Trans-thoracic echocardiography (TTE) is performed in the resting position. Trans-esophageal echocardiography (TEE) is performed under surface anaesthesia with bupivacaine or intravenous anaesthesia. We comprehensively assess the severity of mitral regurgitation according to American Society of Echocardiography (ASE) guideline.
Procedure: TEER — Two commercial cliping systems are available for clinical use: the G3 MitraclipTM and the G4 MitraclipTM (Abbott), DragonflyTM (Dejin), which will be introduced to the Chinese market in 2024, with the specific choice determined by the operator. The patient receives general anaesthesia (intravenous and endotracheal). The operator performs the procedure according to the recommended surgical steps in the product manual, guided by X-ray and trans-esophageal echocardiography. Postoperative MR ≤2+ is considered successful, and if the result is unsatisfactory, 1-2 additional clips are given.

SUMMARY:
To investigate the efficacy and safety of transcatheter mitral valve edge-to-edge repair (TEER) for severe degenerative mitral regurgitation (DMR) patients of low to intermediate surgery risk.

DETAILED DESCRIPTION:
This is a proposed multicentre, prospective cohort study to enrol and follow up severe DMR patients of low to intermediate surgery risk who underwent TEER, and surgical historical controls. The primary efficacy endpoints are all-cause death and cumulative composite event rate of worsening heart failure at 24 months postoperatively, and the primary safety endpoints are death, secondary surgery, and various complications at 30 days postoperatively. The study aims to investigate the efficacy and safety of TEER in surgical low-intermediate-risk patients with severe DMR, and to inform the subsequent clinical application.

ELIGIBILITY:
Inclusion Criteria: the patient fully meets the following criteria.

1. age ≥ 18 years old
2. DMR ≥ grade 3+ according to UCG integrative approach, referring to the following quantitative indicators: 1) effective regurgitant orifice area (EROA) ≥0.3cm^2; 2) regurgitant volume (RVol) ≥45ml; 3) regurgitant fraction (RF) ≥40%.
3. symptomatic heart failure ( New York Heart Association (NYHA) class II-IV ), or asymptomatic heart failure with left ventricular end systolic dimension (LVESd) ≥40mm or ejection fraction (EF) ≤60%, or new-onset atrial fibrillation, or resting pulmonary artery systolic pressure (PASP) >50mmHg.
4. The patient with American Association of Thoracic Surgeons Score (STS) <8 has surgical indications evaluated by cardiac team.
5. The patient has signed an informed consent form and agreed to regular follow-up for at least 1 year.

Exclusion Criteria: the patient meets any of the following criteria.

1. active infective endocarditis especially occurring in the mitral valve area, or mitral valve perforation.
2. rheumatic mitral valve disease, mitral stenosis or mitral valve orifice area < 4mm^2.
3. combined valve lesions requiring surgery, e.g. severe tricuspid regurgitation or aortic valve disease.
4. the present of tumour, thrombus or redundant organisms in the heart chambers.
5. inability to tolerate intraoperative or postoperative antithrombotic (anticoagulant or antiplate) therapy.
6. acute DMR, e.g. DMR caused by acute papillary muscle rupture.
7. Due to the presence of certain anatomical conditions, patient has a low success rate for TEER assessed by the operator and is not appropriate for enrolment. The conditions include but are not limited to the followings: 1) the venous approach is not suitable for operation, such as thrombus in the approach and small vein diameter; 2) severe calcification presents in the flap leaflet clamping area; 3) mitral valve cleft; 4) multiple regurgitant flow, especially in the internal and external union junction area; 5) Barlow disease; 6) leaflet length <7mm; 7) flail gap >10mm; 8) flail width >15mm.
8. severe cardiac insufficiency ( NYHA class IV or lefr ventricular ejection fraction (LVEF) <20% ), end-stage heart failure status ( American College of Cardiology/American Heart Association (ACC/AHA) Stage D), relying on circulation aids or waiting for heart transplantation.
9. proposed implantation of heart failure device such as cardiac resynchronization therapy/cardiac resynchronization therapy defibrillator (CRT/CRT-D) or cardiac contractility modulation (CCM).
10. untreated severe coronary artery stenosis requiring coronary revascularization, or other cardiac macrovascular disease requiring surgery.
11. hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or structural heart disease leading to heart failure other than dilated heart disease.
12. severe pulmonary hypertension ( PASP >70 mmHg), or pulmonary hypertension associated with no-left heart disease, e.g. pulmonary arterial hypertension (PAH) etc.
13. acute myocardial infarction within 4 weeks before operation.
14. acute cerebrovascular accident within 30 days before operation.
15. acute peptic ulcer or upper gastrointestinal bleeding within 3 months before operation.
16. uncontrolled hyperthyroidism.
17. uncontrolled autoimmune connective tissue diseases especially Behcet's disease and systemic lupus erythematosus (SLE).
18. amyloidosis.
19. severe infections, septicaemia.
20. severe hepatic insufficiency, e.g. acute severe hepatitis, decompensated cirrhosis ( Child-Pugh class C)
21. severe renal insufficiency ( chronic kidney disease (CKD) stage 5: estimated glomerular filtration rate (eGFR) < 15 ml/min or dialysis).
22. hypotensive state, shock ( systolic blood pressure < 90mmHg or mean arterial pressure <70 mmHg with tissue hypoperfusion and urine output < 30 ml/h).
23. uncontrolled diseases of the haematological system: acute gastrointestinal bleeding, intracranial haemorrhage or haemorrhage from other organs, acute pulmonary embolism or deep vein thrombosis, congenital or acquired haemorrhagic disease such as haemophilia, anaphylactic purpura and acute leukaemia, severe abnormalities in haematological parameters such as platelet count <20*10^9/L and international normalized ratio (INR) >3.
24. contraindication for TEE, e.g. oesophageal constriction, oesophageal tumour, oesophageal fistula, oesophageal varices, cervical vertebral instability, etc.
25. contraindication for intravenous anaesthesia, e.g. allergy to anaesthetics.
26. pregnancy or breastfeeding.
27. The patient does not sign an informed consent form.
28. expected survival less than 1 year.
29. The patient with poor compliance is not thought to complete follow-up visits.
30. The patient is participating in an experimental drug or other device study with an incomplete primary endpoint, or the patient is participating in an unfinished experimental drug or other device study that would clinically interfere with our study endpoints.
31. Due to other reasons the patient is not suitable for enrollment assessed by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe DMR patients of low to intermediate surgery risk who underwent TEER.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
cumulative composite event rate of the main adverse events | time of operation to 30 days after operation
  The main adverse events: death, acute myocardial infarction, requiring secondary therapy for valve treatment failure, requiring non-scheduled cardiovascular emergency surgery for main complications, stroke, kidney failure, deep infection, >48 hours mechanical ventilation, new-onset atrial fibrillation, deep vein thrombosis, pulmonary embolism, sepsis, haemorrhage, blood transfusion >2U
cumulative composite event rate of all-cause death and worsening heart failure | time of operation to 24 months after operation
  all-cause mortality: deaths from all causes including cardiovascular and non-cardiovascular deaths. worsening heart failure: heart failure rehospitalization, worsening heart failure needing emergency room visit, NYHA classification increased by one, ineffective escalation of medication on outpatient service, receiving intravenous diuretic therapy on outpatient or emergency service.

CONTACTS AND LOCATIONS:
Overall Officials: Yangxin Chen, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided